CLINICAL TRIAL: NCT06968286
Title: The Effect of Locally Dilvered Ciprofloxacine Loaded Injectable Platelet-rich Fibrin as an Adjunct to Non-surgical Periodontal Therapy on the Gingival Crevicular Level of Interleukin 6: A Randomized Controlled Clinical Study
Brief Title: The Effect of Locally Dilvered Ciprofloxacine Loaded Injectable Platelet-rich Fibrin as an Adjunct to Non-surgical Periodontal Therapy on the Gingival Crevicular Level of Interleukin 6
Acronym: PRF & CIP-iPRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Suez canal ethical committee; shaimaa Morsy (Other: Suez Canal university)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis Stage II
Keywords: periodontitis; SRP; i-PRF; ciprofloxacine; IL-6
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: The concentration of the ciprofloxacin drug to be loaded in iPRF will be decided based on the study of Murugan et al., 2024. According to their study, 1 mg/mL of the drug concentration will be found to be biocompatible with maximum efficacy and showed a sustained release of 59% of the loaded drug at the end of the 14-day observation. 1 mg of the drug will be weighed and mixed with 100 μL of deionized water and shaken for 30 seconds to make the drug completely soluble, which will be done just before the blood collection from the participants.
  Preparation of the Drug-loaded i-PRF Then, 900 μL of the obtained i-PRF will be dispensed in a vial containing a 1-mg/100 μL solution of ciprofloxacin and shaken gently for 10 seconds to obtain a homogenous mix with a final concentration of 1 mg/mL.
  Local Delivery of Ciprofloxacin-loaded i-PRF This mixture will further immediately loaded in a 1-mL insulin syringe and injected into the periodontal pocket until it filled the pocket and overflows
Who Masked: Outcomes Assessor
Masking Description: This RCT will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SRP (Active Comparator): prticipants with periodontitis will be treated with conventional periodontal therapy with non surgical scaling and root planning
  Interventions: Procedure: SRP
- SRP+i-PRF (Active Comparator): participants with periodontitis will be treated with nonsurgical periodontal therapy combined with local delivery of injectable platelet rich fibrin
  Interventions: Procedure: SRP+Injectable platelet rich fibrin
- SRP+ciprofloxacine loaded i-PRF (Active Comparator): The concentration of the ciprofloxacin drug to be loaded in iPRF will be decided based on the study of Murugan et al., 2024. According to their study, 1 mg/mL of the drug concentration will be found to be biocompatible with maximum efficacy and showed a sustained release of 59% of the loaded drug at the end of the 14-day observation. 1 mg of the drug will be weighed and mixed with 100 μL of deionized water and shaken for 30 seconds to make the drug completely soluble, which will be done just before the blood collection from the participants.
  Preparation of the Drug-loaded i-PRF Then, 900 μL of the obtained i-PRF will be dispensed in a vial containing a 1-mg/100 μL solution of ciprofloxacin and shaken gently for 10 seconds to obtain a homogenous mix with a final concentration of 1 mg/mL.
  Local Delivery of Ciprofloxacin-loaded i-PRF This mixture will further immediately loaded in a 1-mL insulin syringe and injected into the periodontal pocket until it filled the pocket
  Interventions: Procedure: SRP+ciprofloxacine loaded iPRF

INTERVENTIONS:
Procedure: SRP — participants with periodontitis treated with scaling and root planning
  Arms: SRP
Procedure: SRP+Injectable platelet rich fibrin — The iPRF will be prepared by the same operator according to the protocol developed by Miron and Choukron in 2017. It involves collecting 10 mL of intravenous blood from the participant using venipuncture of the antecubital vein under sterile conditions. The collected blood is transferred to a plain sterile test tube without anticoagulant and immediately subjected to centrifugation at 70-g force at 700 rpm for 3 minutes. After centrifugation, the blood separates into two parts: the bottom layer consists of a red blood cell compartment, and the top layer is platelet-rich fibrin plasma, which is still in liquid consistency. The top platelet-rich fibrin layer is aspirated into a 2-mL syringe and locally delivered in to the periodontal pocket
  Arms: SRP+i-PRF
Procedure: SRP+ciprofloxacine loaded iPRF — The concentration of the ciprofloxacin drug to be loaded in iPRF will be decided based on the study of Murugan et al., 2024. According to their study, 1 mg/mL of the drug concentration will be found to be biocompatible with maximum efficacy and showed a sustained release of 59% of the loaded drug at the end of the 14-day observation. 1 mg of the drug will be weighed and mixed with 100 μL of deionized water and shaken for 30 seconds to make the drug completely soluble, which will be done just before the blood collection from the participants. Then, 900 μL of the obtained i-PRF will be dispensed in a vial containing a 1-mg/100 μL solution of ciprofloxacin and shaken gently for 10 seconds to obtain a homogenous mix with a final concentration of 1 mg/mL.
  This mixture will further immediately loaded in a 1-mL insulin syringe and injected into the periodontal pocket until it filled the pocket
  Arms: SRP+ciprofloxacine loaded i-PRF

SUMMARY:
Sixty periodontally diseased patients will be enrolled in the study. After the patients are randomly divided into one of three treated groups, group 1 (n=20), SRP only; group 2 (n=20), SRP + i-PRF; and group 3 (n=20), P + Cip-loaded i-PRF. Clinical parameters (probing depth [PD], clinical attachment level [CAL], gingival index [GI], plaque index [PI], and level of IL6 in the GCF from baseline to 1 and 3 months of follow-up).

DETAILED DESCRIPTION:
The current randomized, controlled, parallel-design study will be conducted at Suez Canal University's Oral Medicine and Periodontology Department following approval of the study design by the Institutional Review Board and Ethics Committee (931/2024).

Murugan et al. (2024) published a formula that will be used to determine the clinical trial's sample size. According to the following inclusion and exclusion criteria, the study population will be chosen from the subjects who visited the outpatient section of the Department of Oral Medicine and Periodontology Department, Suez Canal University, ion, the sample size was 20 in each group.

Randomization

A computer-generated randomization list utilizing RANDOM.ORG software (www.random.org) with a 1:1 allocation ratio will be used to allocate patients at random to the SRP (control), SRP+I-PRF, or SRP+CIP-loaded I-PRF groups. A non-recruiting faculty member (RA) issued each participant a number, which was then hidden in opaque, sealed envelopes. When adjunctive therapy will be applied, the sealed envelope will be opened to disclose the allocated treatment, and the number will be chosen by the RA for concealment.

Blinding Because it will be unavoidable for the participants and the physician performing the nonsurgical procedure (SH) to be blinded to the interventions, this RCT will be blinded, with the statistician and outcome assessors (MA) blinded.

Patient grouping:

According to the treatment procedure, all 60 selected patients will be randomly allocated to one of the three groups:

Group 1 (n=20): This group will be treated only with SRP without any adjunct therapy.

Group 2 (n=20) After SRP, this group will be treated with the delivery of drug-free i-PRF into the periodontal pocket and gingival tissue adjacent to the pocket. The i-PRF will be applied only once.

Group 3 (n=20): Ciprofloxacin-loaded i-PRF will be administered to this group's periodontal pocket and gingival tissue next to the pocket wall following SRP. Throughout the course of the study, the i-PRF will be used just once.

Preparation of ciprofloxacin solution

Based on the research of Murugan et al., 2024, the ciprofloxacin medication concentration to be loaded in i-PRF will be determined. After a 14-day observation period, their study found that a medication concentration of 1 mg/mL will be biocompatible, have the highest efficacy, and demonstrate a sustained release of 59% of the loaded drug. Just before the participants' blood is drawn, one milligram of the medication will be weighed, combined with 100 μL of deionized water, and shaken for 30 seconds to make the drug fully soluble.

Collection of i-PRF

The i-PRF will be prepared by the same operator using the procedure developed by Miron and Choukron in 2017. This protocol involves obtaining 10 mL of intravenous blood by venipuncturing the participant's antecubital vein under sterile conditions. Immediately after collection, the blood will be centrifuged in a sterile, simple test tube without an anticoagulant for three minutes at 700 rpm and 70 g force. The blood splits into two layers after centrifugation: the top layer is composed of platelet-rich fibrin plasma, which is still liquid, and the bottom layer is composed of a compartment for red blood cells. The top layer of platelet-rich fibrin will be aspirated using a 2-mL syringe and then locally administered into the periodontal pocket for group II.

Preparation of ciprofloxacin-loaded i-PRF

To create a homogeneous mixture with a final concentration of 1 mg/mL, PRF will then be distributed in a vial containing a 1-mg/100 μL solution of ciprofloxacin and gently shaken for 10 seconds. (Murugan1 & Jayakumar 2023)

Local Delivery of Ciprofloxacin-loaded i-PRF

Before it turns into a gel in the group III participants, this combination will also be placed right away into a 1-mL insulin syringe and injected into the periodontal pocket until it fills the pocket and overflows into the tissue next to the periodontal pocket. As previously mentioned, plain i-PRF will be administered to group II participants at the experimental sites. All study participants received postoperative instructions. None of the subjects had a prescription for mouthwash or any other medications, and they will be asked to return for follow-up after one or three weeks.

Clinical assessment

The clinical parameters of the target sites will be measured using a William's probe (Dentsplay, USA) at baseline, 1 month, and 3 months after the treatment. The periodontal parameters included *plaque index (PI) , (Silness & Loe 1964),

To determine the plaque index of the patients, their dental plaque thickness will be evaluated by probing the mesial, distal, buccal, and palatal surfaces of all teeth using a Williams periodontal probe. The plaque index of an individual will be determined by summing the values obtained for each tooth and calculating the averages. To determine the plaque index, Silness & Löe (14) reference values were taken as a basis:

Plaque index 0: No plaque is in the area adjacent to the gingiva. Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.

Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.

Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.

*gingival index (GI),

To determine the gingival index of the patients, gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of all teeth will be evaluated. The gingival index of an individual will be obtained by summing the values determined for each tooth and calculating the averages. To determine the gingival index, Löe & Silness (15) reference values were taken as a basis:

Gingival index 0: Healthy gums. Gingival index 1: Mild discoloration and edematous gingiva. No bleeding on probing.

Gingival index 2: Red, edematous, and shiny gingiva. There is bleeding on probing.

Gingival index 3: Red, edematous, and ulcerated gingiva. There is spontaneous bleeding.

* Pocket depth (PD) (Ramfjord 1967) was assessed from the gingival margin to the base of the pocket,
* Clinical attachment level (CAL) assessed from the cementoenamel junction (CEJ) to the base of the pocket.

Collection of GCF for IL6 detection

GCF samples will be collected from one area from a tooth showing PPD ≤ 5 mm with the highest clinical signs of both inflammation. Supragingival plaque will be removed using a sterile curette without touching the gingival margins, and the area will be gently dried. Cotton rollers were then used to isolate the area in order to avoid contaminating it with saliva. Filter paper (Periopaper, Proflow; Amityville, NY, USA) was used to collect GCF. After carefully inserting paper strips into the gingival sulcus until they encountered only slight resistance, they were left there for 30 seconds. Blood- and saliva-contaminated strips were thrown away. Following the measurement of the GCF volume of each strip using precalibrated electronic impedance equipment (Periotron 8000, ProFlow; Amityville, NY, USA), the strips will be promptly placed into sterile polypropylene tubes and kept at -80°C until analysis.

Each filter paper strip's GCF will be eluted into PBS in the following manner: samples will be kept at 4°C for two hours before the IL-6 tests. After each strip was raised to the eluent's surface, 350 μL of PBS was added, for a total final volume of 600 μL. The samples were then centrifuged for 10 minutes at 10,000 rpm and chilled for an additional 20 minutes at 4°C. The strips will be eventually thrown away.

IL-6 will be analyzed using commercial ELISA kits (R and D Systems, Abingdon, Oxon, UK). A quantitative "sandwich" enzyme immunoassay method is used in the kit. A 96-well microplate will be precoated with an anti-human monoclonal antibody specific to IL-6. In the presence of IL-6, the immobilized antibody bound it. Each well received 200 μL of an enzyme-linked (horseradish peroxidase) polyclonal antibody specific for IL-6 (goat antihuman) following the washing of unattached proteins.

200 μL of a substrate solution will then be added, and the amount of IL-6 that will be bound in the first stage was shown by the color that appeared. Using a microplate reader set to 450 nm with wavelength correction set to 540 nm, the color intensity (optical density) will be determined in 30 minutes. By plotting the concentration of the IL-6 standards (2000, 1000, 500, 250, 125, 62.5, 31.2, and 0 pg/mL) against their optical density, a standard curve was created, and the IL-6 concentration was ascertained. The IL-6 concentration (pg/mL) was then calculated by dividing the amount of IL-6 by the GCF volume (μL), and the pg of IL-6 in each sample (total amount) was computed. The ELISA assays will be performed twice, and the concentrations and total quantities of the cytokine will be determined using the mean values.

ELIGIBILITY:
Inclusion criteria

* The age range of thirty to forty-five
* The participants were diagnosed with stage II grade B periodontitis based on the 2018 classification.
* Participants who have at least two areas with a probing depth (PD) of ≤5 mm and have periodontal disease
* Clinical attachment loss (CAL) values of ≥2 mm or more in participants with periodontal disorders. (Elgendy et al ., 2015)

Exclusion Criteria:

* Pregnant and lactating women
* Use of immunosuppressive medications, consumption of antibiotics, and any antioxidants and anti-inflammatory agents in the last three months
* A history of periodontal therapy in the preceding one year
* Subjects with hemoglobin levels < 11 mg/dL
* Subject participating in any other clinical trials
* Insulin-dependent diabetes

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
change in the clinical attachment level, change in pocket depth | baseline, 1 month and 3 months
  recorded by periodontal probe at baseline, 1 month and 3 months postoperative follow-up interval

SECONDARY OUTCOMES:
detection of concentration of interleukin 6 after nonsurgical periodontal treatment combined with local delivery of iPRF or ciprofloxacine loaded PRF | baseline, 1 month and 3 months
  GCF will be collected at baseline and 1 and 3 months postoperatively using a Periopaper strip (Oraflow, NY, USA). Prior to collection of GCF, the teeth will be isolated by cotton rolls. Then, a gentle water and air spray will be used to eliminate blood and saliva from the test and control teeth. Using a Periopaper strip, GCF will be collected at the mesial and distal sites of the study and control teeth. The PerioPaper strip will be inserted into the sulcus until resistance is felt and remain there for 30 seconds. In case of contamination with blood or saliva, it will be discarded and the procedure will be repeated. After collection of GCF, the periopaper strip will be sealed in sterile polypropylene containers and stored at -80 °C until ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: abdelnasser mohamed elrefaei, professor, Study Director — professor of oral medicine and periodontology
Locations (1):
- Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns, ethical considerations, and/or regulatory restrictions. Additionally, data-sharing agreements or institutional policies may limit the ability to make IPD publicly available."

REFERENCES:
- See also: J Adv Periodontol Implant Dent. 2024 Sep 11;16(2):94-102. doi: 10.34172/japid.2024.021 — https://pmc.ncbi.nlm.nih.gov/articles/PMC11699261/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/39758269/